CLINICAL TRIAL: NCT02735278
Title: Are There Different Objective Fixation Disparity Values for Two Different Test Paradigms: Similar to Reading Dot Presentation and Text Reading? - How This Phenomenon Can be Explained
Brief Title: Are There Different Objective Fixation Disparity Values for Two Different Test Paradigms
Status: Completed | Type: Observational
Sponsor: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Responsible Party: Principal Investigator, Remo Poffa, M.Sc Vision Science (Optometry), University of Applied Sciences and Arts Northwestern Switzerland
Other Study IDs: T426-0034-2
Record Dates: First submitted 2016-03-23; First posted 2016-04-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Vision Disparity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: different test paradigms

SUMMARY:
In optometry, binocular coordination is measured subjectively. The result is subjective fixation disparity. In research different experiments have proven, that subjective and objective fixation disparity are different. A binocular eyetracker has to be calibrated. There are two well known calibration methods: associated and dissociated calibration. Objective fixation disparity is measured in arcMin. Therefore, the precision of the eyetracker plays a crucial role. Now, the investigators try to compare dissociated calibration with polarized filters and associated calibration under different test paradigms.

ELIGIBILITY:
Inclusion Criteria:

* VA without glasses/contact lenses 0.63
* Accurate accommodation on 57cm

Exclusion Criteria:

* Tiredness at day of investigation
* Presbyopia
* Alcohol or drug abuse
* No eye related pathology
* No strabism
* No known epilepsy-attack in family

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adults without binocular problems
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Fixation disparity in arcMin during a reading and reading related dot paradigm | Through study completion, up to 10 months
  With an eyetracker fixation disparity will be measured on an objective way. The scale will be arcMin and test paradigm a reading tast and a dot task, similar to reading.

IPD SHARING:
Plan to Share IPD: No